CLINICAL TRIAL: NCT04928703
Title: A Phase 0, Double-Blind, Randomized, Placebo-Controlled, Crossover Study to Assess Ketamine-induced Changes in ERP Biomarkers in Healthy Volunteers
Brief Title: Effects of Ketamine on ERP/EEG Measures in Healthy Volunteers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: ERP Biomarker Qualification Consortium (Industry)
Collaborators: Alkermes, Inc. (Industry); Anavex Life Sciences Corp. (Industry); Astellas Pharma Inc (Industry); H. Lundbeck A/S (Industry); Merck Sharp & Dohme LLC (Industry); Novartis (Industry); Sage Therapeutics (Industry); Takeda (Industry); Apex Innovative Sciences (Unknown); COGNISION (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: EBS-B
Record Dates: First submitted 2021-05-28; First posted 2021-06-16 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Healthy
Keywords: Event-related potential; Electroencephalogram; ERP; EEG; Ketamine; Mismatch Negativity; MMN; N100; P3a; P3b; P300
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: Single Dose, Placebo-Controlled, 3-Arm Crossover
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): Visit 2: Placebo - Placebo; Visit 3: Placebo - Ketamine; Visit 4: Placebo - Ketamine
  Interventions: Drug: Ketamine
- Arm 2 (Experimental): Visit 2: Placebo - Ketamine; Visit 3: Placebo - Placebo; Visit 4: Placebo - Ketamine
  Interventions: Drug: Ketamine
- Arm 3 (Experimental): Visit 2: Placebo - Ketamine; Visit 3: Placebo - Ketamine; Visit 4: Placebo - Placebo
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Ketamine IV administration

SUMMARY:
This is a Phase 0, Double-Blind, Randomized, Placebo-Controlled, Crossover Study to assess the changes in ERP Biomarkers in Healthy Volunteers before and after administration of a sub-anesthetic dose of ketamine. Primary objectives are to quantify the effect size of ketamine-induced changes on MMN from a duration-deviant auditory oddball ERP test and to quantify the variability of ketamine-induced changes on MMN from a duration-deviant auditory oddball ERP test.

DETAILED DESCRIPTION:
The effects of ketamine and similar compounds on brain function have become of significant interest to pharma companies in the past few years. These effects are often used as a model for the glutamatergic hypofunction hypothesis of schizophrenia and therefore drugs targeting schizophrenia are being trialed to reverse or block the effects of ketamine. Esketamine has been recently approved as a potent treatment for depression so many pharma companies are trying to leverage ketamine-like modulation of the NMDA receptors as novel targets for depression.

This heightened focus on NMDAr modulators has lead industry and academia to advance methods to measure these effects. Many studies have been performed using EEG and ERP techniques to measure the effect on brain function of ketamine administration but no study has been performed, to our knowledge, that has attempted to measure the variability and reproducibility of these effects. Furthermore, there is some evidence from the scientific literature and from unpublished results from industry-sponsored studies that ketamine may have a disordinal effect on various electrophysiologic measures, particularly the amplitude of the mismatch negativity (MMN) from an auditory oddball ERP test.

In this study we will run various EEG/ERP tests on participants during a placebo administration and during two ketamine administrations separated by washout periods. This will allow, for the first time, the evaluation of the test-retest variability of a range ERP/EEG measures under ketamine administration vs placebo. This may also allow us to test the hypothesis that ketamine has a disordinal effect on different subjects and this disordinality can be predicted from a baseline (placebo) measurement.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects 21-40 years of age, inclusive at Visit 1 (Screening).
2. Female subjects with a negative serum pregnancy test prior to entry into the study and who are practicing an adequate method of birth control (e.g., oral or parenteral contraceptives, intrauterine device, barrier, abstinence) and who do not plan to become pregnant during the study and for 30 days after the last dose of ketamine.
3. Ability to understand the requirements of the study, provide written informed consent, abide by the study restrictions, and agree to return for the required assessments.
4. Subject is judged to be in good health as determined by the investigator.
5. Body mass index (BMI ) between 18.5 and 30.0 (inclusive) at Visit 1 (Screening).
6. Ability to detect a 1000 and 2000 Hz tone at 40 dB in both ears, at Visit 1 (Screening).
7. Ability to tolerate the electrode cap for the duration of the testing session.

Exclusion Criteria:

1. Clinically significant alcohol or other substance abuse within the last 1 year, in the opinion of the investigator; or unable to abstain from alcoholic beverages during the course of the study.
2. Positive alcohol/drug screen for drugs of abuse (with the exception of a positive result considered by the investigator to be directly attributable to prescription medication approved for subject use) such as phencyclidine, benzodiazepines, opiates, cocaine, cannabinoids, amphetamines, and cotinine at any Visit.
3. Excessive caffeine use (defined as habitual consumption of > 400 mg caffeine per day [~ four 8 oz. cups brewed caffeinated coffee or tea, ~ ten 12 oz. cans caffeinated soda or ~ two "energy shot" drinks]), or unable to abstain from caffeine on Visits 2-4.
4. Use of products containing nicotine (tobacco or vaping products) 60 minutes prior to dosing on Visits 2-4.
5. Current or prior history (defined as in the past 6 months) of treatment with N-methyl-D-aspartate receptor (NMDAR) ligands including ketamine, amantadine, dextromethorphan, memantine, methadone, dextropropoxyphene, or ketobemidone.
6. History of allergy, sensitivity, or intolerance to NMDAR ligands including ketamine, amantadine, dextromethorphan, memantine, methadone, dextropropoxyphene, or ketobemidone.
7. Any impairment, activity, or situation that in the judgment of the investigator would prevent satisfactory completion of the study protocol.
8. History of significant psychiatric, neurologic (e.g. Huntington's, Parkinson's, Alzheimer's, Multiple Sclerosis, Type I or Type II diabetes mellitus, or a history of seizures, epilepsy, or strokes), or cognitive disorders (e.g. bipolar, schizophrenia, psychosis), or current (within 12 months prior to screening) psychiatric or cognitive disorders such as major depression, suicidal ideation, dementia, or anxiety disorders).
9. Abnormal medical history, or concurrent conditions that, in the opinion of the investigator or sponsor designated medical monitor, would preclude safe study participation, or interfere with study procedures/assessments.
10. History of severe renal or hepatic impairment, in the opinion of the investigator or the sponsor medical monitor.
11. Known history of significant cardiovascular condition such as myocardial infarction, congestive heart failure, clinically significant arrhythmias, current uncontrolled cardiac arrhythmias, angina, acute ischemia.
12. Hypertension characterized by resting systolic blood pressure > 140 mmHg or resting diastolic > 90 mmHg or tachycardia defined as a resting HR ≥ 120 bpm or bradycardia defined as a resting HR of ≤ 50 bpm, at any Visit.
13. Hypotension with an abnormal supine blood pressure defined as SBP < 90 mmHg or DBP <60 mmHg at any Visit.
14. Orthostatic hypotension consisting of a SBP change of ≥ 30 mmHg or a DBP change of ≥ 20 mmHg at 3 minutes after standing from a supine position at any Visit.
15. Resting heart rate < 45 or > 95 beats per minute.
16. A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms) or any other relevant ECG finding at Visit 1 (Screening).
17. A history of additional risk factors for Torsade de Pointes (such as heart failure, hypokalaemia, or family history of Long QT Syndrome).
18. Current evidence of dysplasia or history of malignancy (including lymphoma and leukemia) in the last 5 years, with the exception of successfully treated non-metastatic basal cell or squamous cell carcinoma of the skin or localized carcinoma in situ of the cervix.
19. Human immunodeficiency virus (HIV) infection, hepatitis, or other ongoing infectious disease that the investigator considers clinically significant.
20. History of gastrointestinal disease or surgery (except simple appendectomy or hernia repair), which can influence the absorption of the study drug.
21. Evidence of an infection at the time of clinic admission, in the opinion of the investigator.
22. Received an investigational product or device within 30 days (or 5 half-lives, whichever is longer) of dosing.
23. Use of first generation, sedating H1 antihistamines or sedative-hypnotic medications within 1 week prior to dosing.
24. Poor venous access; or have donated or had a significant loss of blood or plasma within 8 weeks of dosing.
25. Known allergy to latex.
26. Prior adverse reaction to ketamine or esketamine.
27. Medical history, conditions, or situations that, in the opinion of the investigator, would preclude safe study participation, or interfere with study procedures/assessments.
28. In addition to these criteria, the investigator may discontinue subjects at any time based on his or her clinical judgment.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2022-05-26 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
Ketamine-induced changes in Amplitude for parameters from the ERP tests. | Pre-intervention/Dosing
  Amplitude changes (in microvolts) for the following parameters from the ERP tests:
  1. Passive, Duration-deviant, Oddball ERP
  a. MMN

SECONDARY OUTCOMES:
Ketamine-induced changes in Amplitude for parameters from the ERP tests. | Pre-intervention/Dosing
  Amplitude changes (in microvolts) for the following parameters from the ERP tests:
  1. Passive, Duration-deviant, Oddball ERP
     1. N100
     2. P3a
  2. Active, Auditory Oddball ERP
     1. N100
     2. N200
     3. P3b
Ketamine-induced changes in Latency for parameters from the ERP tests. | Pre-intervention/Dosing
  Latency changes (in milliseconds) for the following parameters from the ERP tests:
  1. Passive, Duration-deviant, Oddball ERP
     1. N100
     2. MMN
     3. P3a
  2. Active, Auditory Oddball ERP
     1. N100
     2. N200
     3. P3b
Ketamine-induced change in Task Accuracy from the behavioral response during the active, auditory oddball ERP test. | Pre-intervention/Dosing
  Change in Task Accuracy as a percentage of correct behavioral responses during the active, auditory oddball ERP test.
Ketamine-induced change in Reaction Time from the behavioral response during the active, auditory oddball ERP test. | Pre-intervention/Dosing
  Change in Reaction Time for the correct behavioral responses measured in milliseconds during the active, auditory oddball ERP test.
Ketamine-induced change in Evoked Power from the auditory steady-state response (ASSR) paradigm. | Pre-intervention/Dosing
  Change in Evoked Power measured in µv2/Hz from the ASSR paradigm.
Ketamine-induced change in Inter-trial coherence (ITC) from the auditory steady-state response (ASSR) paradigm. | Pre-intervention/Dosing
  Inter-trial coherence (ITC) from the ASSR paradigm will be measured on a scale between 0 (no coherence) and 1 (maximum coherence). Outcome measure will be change in ITC.
Ketamine-induced changes in Absolute Power for Pharmaco-EEG parameters per IPEG guidelines. | Pre-intervention/Dosing
  Changes in Absolute Power (measured in µv2/Hz) for the following Pharmaco-EEG parameters:
  * Delta power
  * Theta power
  * Alpha power
  * Beta power
  * Gamma power
  * Total power
Ketamine-induced changes in Relative Power for Pharmaco-EEG parameters per IPEG guidelines. | Pre-intervention/Dosing
  Relative Power for Pharmaco-EEG parameters will be measured on a scale from 0 (no power in frequency band) to 1 (all EEG power in that frequency band). Outcome measures will be changes in Relative Power for the following Pharmaco-EEG parameters:
  * Delta power
  * Theta power
  * Alpha power
  * Beta power
Ketamine-induced change in the Dominant Frequency for the Alpha frequency band per IPEG guidelines. | Pre-intervention/Dosing
  Dominant frequency will be measured in Hz in the frequency interval between 6.0 and < 12.5 Hz. Outcome measure will be change in the Dominant Frequency for the Alpha frequency band.
Ketamine-induced changes in Slow Wave Index per IPEG guidelines. | Pre-intervention/Dosing
  Slow Wave Index (SWI) will be calculated as Alpha/(Delta+Theta), and will be measured as ratio. Outcome measure will be change in SWI.
Ketamine-induced changes in Theta/Beta ratio per IPEG guidelines. | Pre-intervention/Dosing
  Theta/Beta (TBR) will be measured as ratio. Outcome measure will be change in TBR.
Correlations between Ketamine blood concentration and Ketamine-induced changes in Amplitude for parameters from the ERP tests. | Pre-intervention/Dosing
  Correlations between ketamine blood concentration and amplitude changes (in microvolts) for the following parameters from the ERP tests:
  1. Passive, Duration-deviant, Oddball ERP
     a. MMN
  2. Passive, Duration-deviant, Oddball ERP
     1. N100
     2. P3a
  3. Active, Auditory Oddball ERP
     1. N100
     2. N200
     3. P3b
Correlations between Ketamine blood concentration and Ketamine-induced changes in Latency for parameters from the ERP tests. | Pre-intervention/Dosing
  Correlations between ketamine blood concentration and latency changes (in milliseconds) for the following parameters from the ERP tests:
  1. Passive, Duration-deviant, Oddball ERP
     a. MMN
  2. Passive, Duration-deviant, Oddball ERP
     1. N100
     2. P3a
  3. Active, Auditory Oddball ERP
     1. N100
     2. N200
     3. P3b
Correlation between Ketamine blood concentration and Ketamine-induced change in Task Accuracy from the behavioral response during the active, auditory oddball ERP test. | Pre-intervention/Dosing
  Correlation between Ketamine blood concentration and change in Task Accuracy measured as a percentage of correct behavioral responses during the active, auditory oddball ERP test.
Correlation between Ketamine blood concentration and Ketamine-induced change in Reaction Time from the behavioral response during the active, auditory oddball ERP test. | Pre-intervention/Dosing
  Correlation between Ketamine blood concentration and change in Reaction Time for the correct behavioral responses measured in milliseconds during the active, auditory oddball ERP test.
Correlation between Ketamine blood concentration and Ketamine-induced change in Evoked Power from the auditory steady-state response (ASSR) paradigm. | Pre-intervention/Dosing
  Correlation between Ketamine blood concentration and change in Evoked Power measured in µv2/Hz from the ASSR paradigm.
Correlation between Ketamine blood concentration and Ketamine-induced change in Inter-trial coherence (ITC) from the auditory steady-state response (ASSR) paradigm. | Pre-intervention/Dosing
  Correlation between Ketamine blood concentration and change in Inter-trial coherence (ITC) from the ASSR paradigm. Change in ITC will be measured on a scale between 0 (no coherence) and 1 (maximum coherence).
Correlation between Ketamine blood concentration and Ketamine-induced changes in Absolute Power for Pharmaco-EEG parameters. | Pre-intervention/Dosing
  Correlation between Ketamine blood concentration and changes in Absolute Power (measured in µv2/Hz) for the following Pharmaco-EEG parameters:
  * Delta power
  * Theta power
  * Alpha power
  * Beta power
  * Gamma power
  * Total power
Correlation between Ketamine blood concentration and Ketamine-induced changes in Relative Power for Pharmaco-EEG parameters. | Pre-intervention/Dosing
  Correlation between Ketamine blood concentration and changes in Relative Power for the following Pharmaco-EEG parameters:
  * Delta power
  * Theta power
  * Alpha power
  * Beta power
Correlation between Ketamine blood concentration and Ketamine-induced change in the Dominant Frequency for the Alpha frequency band. | Pre-intervention/Dosing
  Correlation between Ketamine blood concentration and Dominant frequency for the Alpha frequency band measured in Hz in the frequency interval between 6.0 and < 12.5 Hz.
Correlation between Ketamine blood concentration and Ketamine-induced changes in Slow Wave Index. | Pre-intervention/Dosing
  Correlation between Ketamine blood concentration and changes Slow Wave Index (SWI) calculated as Alpha/(Delta+Theta) ratio.
Correlation between Ketamine blood concentration and Ketamine-induced changes in Theta/Beta ratio. | Pre-intervention/Dosing
  Correlation between Ketamine blood concentration and changes in Theta/Beta ratio (TBR).

CONTACTS AND LOCATIONS:
Overall Officials: Marco Cecchi, PhD, Principal Investigator — The ERP Biomarker Qualification Consortium
Locations (1):
- Hassman Research Institute, Marlton, New Jersey, United States